CLINICAL TRIAL: NCT06541535
Title: Comparison of Saline and Ringer Lactate in Patients With Severe Diabetic Ketoacidosis (DRINK) : a Double-blind Randomized Controlled Trial
Brief Title: Fluid Administration in Ketoacidosis (DRINK)
Acronym: DRINK
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-API-03
Record Dates: First submitted 2024-07-08; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Keto-acidosis
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isotonic saline (Active Comparator)
  Interventions: Drug: Fluid resuscitation with isotonic saline only
- Ringer Lactate (Experimental)
  Interventions: Drug: Fluid resuscitation with Ringer Lactate

INTERVENTIONS:
Drug: Fluid resuscitation with isotonic saline only — Isotonic saline only will be used for fluid resuscitation in the first 48 hours of treatment, according to the protocol of English guidelines:
  * During the first hour of treatment:
    * In the event of systolic arterial hypotension (SAP<90mmHg): administration of 500 mL over 15 minutes, renewable once, then administration of 1L over 1 hour.
    * In the absence of systolic arterial hypotension (SAP>90mmHg): administration of 1L over 1 hour.
  * Between 60 minutes and 8 hours of treatment :
    * 1L over 2 hours, repeated once, then 1L over 4 hours
    * Adjust fluid resuscitation according to clinical tolerance
  * After the first 8 hours:
    * 1L over 4h then 1L over 6h
    * Clinical re-evaluation according to standard of care in participating centers
  Arms: Isotonic saline
Drug: Fluid resuscitation with Ringer Lactate — Ringer Lactate only will be used for fluid resuscitation in the first 48 hours of treatment, according to the protocol of English guidelines:
  * During the first hour of treatment:
    * In the event of systolic arterial hypotension (SAP<90mmHg): administration of 500 mL over 15 minutes, renewable once, then administration of 1L over 1 hour.
    * In the absence of systolic arterial hypotension (SAP>90mmHg): administration of 1L over 1 hour.
  * Between 60 minutes and 8 hours of treatment :
    * 1L over 2 hours, repeated once, then 1L over 4 hours
    * Adjust fluid resuscitation according to clinical tolerance
  * After the first 8 hours:
    * 1L over 4h then 1L over 6h
    * Clinical re-evaluation according to standard of care in participating centers
  Arms: Ringer Lactate

SUMMARY:
Management of severe diabetic ketoacidosis is based on insulin therapy, correction of metabolic disorders and fluid resuscitation. Current recommendations recommend the first-line use of isotonic saline, whose composition is unbalanced, rich in chloride and sodium compared with plasma. Administration of large volumes of isotonic saline is associated with a risk of hyperchloremic metabolic acidosis and acute renal failure. Balanced solutions (e.g. Ringer Lactate) are solutions with a more balanced electrolyte composition close to that of plasma. They could therefore enable diabetic ketoacidosis to be resolved more quickly than isotonic saline, due to a lower risk of hyperchloremic acidosis. Preliminary data suggest a potential benefit of balanced solutions for fluid resuscitation of patients with severe diabetic ketoacidosis in terms of resolution of diabetic ketoacidosis, but no randomized controlled double-blind study to date has compared balanced solution vs. isotonic saline in this context.

ELIGIBILITY:
Inclusion Criteria:

* Admission to emergency department or direct admission to ICU
* Diagnosis of severe diabetic ketoacidosis requiring all the following criteria:
* Blood or capillary glucose > 11 mmol/L
* Ketonemia or ketonuria > 0
* Venous or arterial pH < 7.30 or venous or arterial bicarbonate < 15 mmol/L
* Volume of fluid administered before inclusion <1L

Exclusion Criteria:

* Patients <18 years
* Pregnant women
* Patients under protection
* Patients with a decision to withdraw life-sustaining therapy
* Contraindication to isotonic saline or Ringer Lactate
* Non-affiliation to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Resolution of diabetic ketoacidosis | at 24 hours
  Compare fluid resuscitaiton with Ringer Lactate to isotonic saline on the resolution of diabetic ketoacidosis at 24 hours from admission to Intensive Care Unit (ICU) in patients with severe diabetic ketoacidosis.
  Resolution of ketoacidosis allowing discharge from ICU, defined as the proportion of patients with the following three criteria at 24 hours from ICU admission :
  1. capillary or blood glucose < 11 mmol/L
  2. undetectable ketonemia or ketonuria
  3. venous or arterial pH > 7.35 or venous or arterial bicarbonate > 20 mmol/L

SECONDARY OUTCOMES:
Speed of resolution of metabolic disorders | at 48 hours
  Compare fluid resuscitation with Ringer Lactate and isotonic saline solution on the speed of resolution of metabolic disorders in patients admitted to ICU for severe diabetic ketoacidosis.
  Proportion of patients and number of hours ("Resolution free hours") within 48 hours of ICU admission with the following three criteria:
  1. capillary or blood glucose < 11 mmol/L
  2. undetectable ketonemia or ketonuria
  3. venous or arterial pH > 7.35 or venous or arterial bicarbonate > 20 mmol/L
Time of resolution of metabolic disorders | at 48 hours
  Compare fluid resuscitation with Ringer Lactate and isotonic saline solution on the speed of resolution of metabolic disorders in patients admitted to ICU for severe diabetic ketoacidosis.
  Time (in hours) from ICU admission to obtain one of the following three criteria:
  1. capillary or blood glucose < 11 mmol/L for at least 4 consecutive hours
  2. undetectable ketonemia or ketonuria
  3. venous or arterial pH > 7.35 or venous or arterial bicarbonate > 20 mmol/L
Assess the metabolic tolerance of Ringer Lactate compared to isotonic saline solution | through the end of study average 24 months
  Assess the metabolic tolerance of Ringer Lactate compared to isotonic saline solution in patients admitted to ICU for severe diabetic ketoacidosis.
  Occurrence of serious metabolic disorders during ICU stay, defined as :
  1. Kalemia < 3 mmol/L
  2. Natremia > 145 mmol/L
  3. Chloremia > 110 mmol/L
  4. Phosphoremia < 0.70 mmol/L
  5. Blood glucose < 3.8 mmol/L (i.e. 0.80 g/L)
  6. Persistent ketonemia/ketonuria 24 hours after ICU admission 2. Nature and volume (in liters) of fluid administered before inclusion and during the study period in each group 3. Protocol compliance (expressed as % of volume administered in each group)
Assess the impact of Ringer lactate compared with isotonic saline on renal, neurological and cardiac complications | at 28 days
  To assess the impact of Ringer lactate compared with isotonic saline on renal, neurological and cardiac complications during ICU stay and outcomes of patients admitted to ICU for severe diabetic ketoacidosis.
  Occurrence of adverse events during ICU stay, defined as :
  1. Neurological disorders (Glasgow score)
  2. Acute renal failure (KDIGO classification)
  3. Cardiac disorders (supraventricular and ventricular rhythm disorders, acute coronary syndrome) 2. ICU and hospital length of stay 3. ICU mortality and Day-28 mortality
Assess the impact of Ringer lactate compared with isotonic saline on cardiac complications | at 28 days
  To assess the impact of Ringer lactate compared with isotonic saline on cardiac complications during ICU stay and outcomes of patients admitted to ICU for severe diabetic ketoacidosis.
  Occurrence of adverse events during ICU stay, defined as :
  * Cardiac disorders (supraventricular and ventricular rhythm disorders, acute coronary syndrome)
  * ICU and hospital length of stay
  * ICU mortality and Day-28 mortality
Assess the impact of Ringer lactate compared with isotonic saline on renal complications | at 28 days
  To assess the impact of Ringer lactate compared with isotonic saline on renal, complications during ICU stay and outcomes of patients admitted to ICU for severe diabetic ketoacidosis.
  Measure acute renal failure with KDIGO classification.
  The Kidney Disease: Improving Global Outcomes (KDIGO) classification system stratifies acute kidney injury (AKI) into levels of severity, determined by changes in serum creatinine (SCr) / estimated creatinine clearance (eCCl), as well as changes in urine output. The strata of severity of AKI can be reached by meeting the criteria for changes in SCr / eCCl or changes in urine output. There are three levels of severity, with level 1 being the least severe and level 3 the most severe.
  No cut-off for the study
Assess the impact of Ringer lactate compared with isotonic saline on neurological complications | at 28 days
  To assess the impact of Ringer lactate compared with isotonic saline on neurological complications during ICU stay and outcomes of patients admitted to ICU for severe diabetic ketoacidosis.
  Measure Neurological disorders with Glasgow score. The Glasgow Coma Scale (GCS) is used to objectively describe the extent of impaired consciousness in all types of patients. The scale rates patients on three aspects of reactivity: eye opening, motor responses and verbal responses. It ranges from 3 (coma) to 15 (no disturbance of consciousness). No cut-off for the study.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, France